CLINICAL TRIAL: NCT07035769
Title: A Phase 1, First-in-human, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of Debio 1453P in Healthy Adults
Brief Title: A First-in-Human Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single and Multiple Oral Doses of Debio 1453P in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Wellcome Trust (Other); Germany's Federal Ministry of Research, Technology and Space (BMFTR) (Unknown); Global Antimicrobial Resistance Innovation Fund-(GAMRIF) (Unknown); Novo Nordisk Foundation (NNF) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Debio 1453-101; 2024-519328-26 (Other: EU CT Number); U1111-1315-2035 (Other: WHO Universal Trial Number); 75A50122C00028 (Other Grant/Funding Number: HHS/BARDA OTA Number); 224842/Z/21/Z (Other Grant/Funding Number: Wellcome Trust); NNF23SA0088536 (Other: Novo Nordisk Foundation (NNF)); Agreement Dated 1/30/2023 (Other: Germany's Federal Ministry of Research, Technology and Space (BMFTR)); Agreement Dated 2/28/2023 (Other: Global Antimicrobial Resistance Innovation Fund (GAMRIF))
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Single ascending dose (SAD) (Experimental): Participants will receive a single oral dose of Debio 1453P or placebo in a sequential manner on Day 1.
  Interventions: Drug: Debio 1453P; Drug: Placebo
- Part 2: Multiple ascending dose (MAD) (Experimental): Participants will receive multiple oral doses of Debio 1453P or placebo from Day 1 to Day 5. Debio 1453P initial dose in this part will be based on available data from SAD part.
  Interventions: Drug: Debio 1453P; Drug: Placebo

INTERVENTIONS:
Drug: Debio 1453P — Powder for oral solution
Drug: Placebo — Oral solution

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) of Debio 1453P compared to placebo across different dose levels in healthy adults after single and repeated oral dosing.

ELIGIBILITY:
Inclusion Criteria

1. Signed and dated written informed consent obtained before undertaking any trial-specific procedures.
2. Be within the age range of 18 to 55 years, inclusive, at the time of screening.
3. Have a body mass index (BMI) ≥18.5 and ≤30.0 kg/m^2.

Exclusion criteria

1. History and/or physical examination evidence of any clinically significant disease or disorder, such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal, endocrine, immunological, psychiatric or mental disease or disorder, or mental or legal incapacitation, which, in the opinion of the Investigator, may either put the participant at risk for taking part in the trial, influence the results of the trial, influence the participant's ability to take part in the trial.
2. Any medication (including vaccines, over the counter (OTC) and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements, and hormonal replacement therapy for postmenopausal participants) for 2 weeks or 5 half-lives of the drug, whichever is longer, prior to first administration of trial drug (except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks).
3. History of chronic drug or alcohol abuse (defined as an average intake of more than 21 units of alcohol per week for males and 14 for females. 1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits) in the last 2 years.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs) | Up to 15 months

SECONDARY OUTCOMES:
Plasma Concentration of Debio 1453P | Pre-dose and at multiple timepoints post-dose up to Day 12
  The PK of Debio 1453P will be evaluated in plasma.
Urine Concentration of Debio 1453P | Pre-dose and at multiple timepoints post-dose up to Day 12
  The PK of Debio 1453P will be evaluated in urine.

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Belgium NV - Clinical Pharmacology Unit, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No